#### Viiv Healthcare group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a non-randomized, sequential, fixed-sequence evaluation of prototype dolutegravir liquid formulations versus 5mg dolutegravir dispersible tablets following single-dose fasted-state administrations to normal healthy adult participants

Compound Number : GSK1349572

Effective Date : 17-Apr-2019

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209354.
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Author | Date |
|---|---|
| PPD | 17 Apr 2010 |
| Senior Statistician (Infectious Diseases, Clinical Statistics) | 17-Apr-2019. |

Copyright 2019 the ViiV Healthcare group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Review Confirmations (Method: E-mail):**

| Reviewer | Date |
|------------------------------------------------------------|-------------|
| PPD | |
| Programming Manager (Infectious Diseases, Clinical | 14-Apr-2019 |
| Programming) | |
| PPD | |
| Global Clinical Development Director (Infectious Diseases, | 12-Apr-2019 |
| R&D PCPS GCSD) | |
| , FCP MSc | |
| Director (Clinical Development, Research and Development, | 12-Apr-2019 |
| ViiV Healthcare) | |
| PPD | 12 Apr 2010 |
| Director (Clinical Pharmacology, ViiV Healthcare) | 12-Apr-2019 |
| PPD | 15 Apr 2010 |
| Director (Clinical Pharmacology Modelling and Simulation) | 15-Apr-2019 |
| PPD | 15-Apr-2019 |
| Principal Statistician (Dolutegravir Statistics) | 13-Api-2019 |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignature and Email):

| Approver | Date |
|---|---|
| Statistics Director (Infectious Diseases, Clinical Statistics) [pharma TMF e-Signature] | 17-Apr-2019 |
| Programming Director (Infectious Diseases, Clinical Programming) [email approval] | 16-Apr-2019 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s). Study Design Statistical Hypotheses. | 5<br>5 |
| 3. | PLANI<br>3.1.<br>3.2. | INED ANALYSES Interim Analyses Final Analyses | 8 |
| 4. | ANAL`<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING VENTIONS | 10<br>10 |
| 6. | STUD<br>6.1.<br>6.2. | OY POPULATION ANALYSESOverview of Planned Study Population Analyses | 12 |
| 7. | SAFE <sup>7</sup> .1. 7.2. 7.3. | Adverse Events Analyses 7.1.1. Details of Planned Adverse Event Summaries Clinical Laboratory Analyses 7.2.1. Details of Planned Laboratory Summaries Other Safety Analyses | 14<br>15<br>15 |
| 8. | PHAR<br>8.1. | Primary Pharmacokinetic Analyses | 171717171718181819 |
| | | 8.2.1.1. Drug Concentration Measures | |

## CONFIDENTIAL

| 20035 |
|-------|

| | | 8.2.2. | Summary Measure | 20 |
|---|---|---|---|---|
| | | 8.2.3. | Population of Interest | |
| | | 8.2.4. | Strategy for Intercurrent (Post-Randomization) Events | 21 |
| | | 8.2.5. | Statistical Analyses / Methods | |
| | | | 8.2.5.1. Statistical Methodology Specification | 21 |
| | | 8.2.6. | Details of Planned Pharmacokinetic Displays | 21 |
| ^ | DEEE | DENOGO | | 00 |
| 9. | KEFEI | RENCES | | 23 |
| 10. | APPEI | NDICES. | | 24 |
| | 10.1. | | x 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | 24 |
| | 10.2. | Appendi | x 2: Schedule of Activities | 25 |
| | | 10.2.1. | | |
| | | | 10.2.1.1. Screening Assessments | |
| | | | 10.2.1.2. Treatment Period Assessments | |
| | 10.3. | Appendi | x 3: Study Phases and Treatment Emergent Adverse | |
| | | | | 27 |
| | | 10.3.1. | | |
| | | | 10.3.1.1. Study Phases for Concomitant Medication | |
| | | 10.3.2. | Treatment Emergent Flag for Adverse Events | |
| | 10.4. | | x 4: Data Display Standards & Handling Conventions | |
| | 10.1. | 10.4.1. | Reporting Process | 20 |
| | | 10.4.1. | | |
| | | 10.4.3. | | |
| | 10.5. | | x 5: Derived and Transformed Data | |
| | 10.0. | | General | |
| | | 10.5.1. | | |
| | 10.6. | | x 6: Reporting Standards for Missing Data | |
| | 10.0. | 10.6.1. | | |
| | | 10.6.1. | Handling of Missing Data | |
| | | 10.0.2. | 10.6.2.1. Handling of Missing and Partial Dates | |
| | 10.7. | Annandi | x 7: Values of Potential Clinical Importance | |
| | 10.7. | | x 8: Abbreviations & Trade Marks | |
| | 10.6. | | | |
| | | | Abbreviations | |
| | 10.0 | | Trademarks | |
| | 10.9. | | x 9: List of Data Displays | |
| | | 10.9.1. | Data Display Numbering | |
| | | 10.9.2. | Mock Example Shell Referencing | |
| | | 10.9.3. | Deliverables | |
| | | 10.9.4. | Study Population Tables | |
| | | 10.9.5. | Safety Tables | |
| | | 10.9.6. | Pharmacokinetic Tables | |
| | | 10.9.7. | Pharmacokinetic Figures | |
| | | 10.9.8. | ICH Listings | |
| | 10.10. | Appendi | x 10: Example Mock Shells for Data Displays | 48 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2018N379348_00 | 29-Oct-2018 | Original |
| 2018N379348_01 | 27-Feb-2019 | The original protocol was written assuming that a greater number of prototype formulations would possibly have been tested in the study. Pre-clinical testing yielded only 2 prototypes suitable to take forward clinically. This amendment clarifies the study design for only 2 test formulations. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 01 [(Dated: 27/Feb/2019)].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the relative bioavailability of equivalent doses of single dose prototype liquid formulations containing 10mg equivalent DTG compared to a single dose of 2 x 5mg dispersible DTG tablet dispersed in water. Secondary Objectives To characterize the pharmacokinetics of equivalent doses of a single dose of prototype liquid formulations containing 10mg equivalent DTG and a single dose of 2 x 5mg dispersible DTG tablet dispersed in water. | $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ |
| T | of each formulation |
| To assess the safety and tolerability from single-dose administration of prototype liquid formulations containing 10mg equivalent DTG in healthy participants in a fasted state. | Safety and tolerability parameters as assessed by change from baseline in vital signs (BP and HR), number of participants with adverse events and toxicity grading of clinical laboratory tests. |

BP = Blood Pressure

HR = Heart rate

AUC<sub>(0-t)</sub> = area under the plasma concentration time curve from time zero to the last quantifiable time point

 $AUC_{(0-\infty)}$  = area under the plasma concentration time curve from time zero to infinity

 $AUC_{(0-24)}$  = area under the plasma concentration time curve from time zero to 24 hours

%AUCex=% of AUC(0-∞) that was extrapolated

C<sub>max</sub> = maximum observed concentration

t<sub>max</sub> = time of maximum observed concentration

 $C_{24}$  = concentration at 24h post-dose

Ct = last quantifiable concentration

PK = Pharmacokinetic

t = time of last quantifiable concentration

t<sub>lag</sub> = absorption lag time

λz=apparent elimination rate constant

t<sub>1/2</sub> = the elimination half-life

CL/F = apparent oral clearance

Vz/F= apparent oral volume of distribution

## 2.3. Study Design



# 2.4. Statistical Hypotheses

This study is designed to estimate the relative bioavailability of two experimental liquid formulations of DTG relative to DTG dispersible tablets dispersed in water and dosed in the fasted state.

No formal hypotheses will be tested.

For each pharmacokinetic endpoint (except  $t_{max}$  and  $t_{lag}$ ), point estimates of the geometric mean of each prototype treatment and Reference Treatment are estimated. The ratio of the two estimates (GMR),  $\mu$  (prototype)/ $\mu$  (reference), and its corresponding 90% confidence interval will be constructed.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

There will be no formal interim analyses.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. The study has a non-randomised open label design; however, for internal study reporting, subjects will be assigned randomisation numbers. Therefore, the formal process for unblinding the randomization codes is required.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population Definition / Criteria | | Analyses Evaluated |
|---|---|---|
| Screened | All participants who sign the ICF | Screen Failures |
| Enrolled | <ul> <li>All participants who passed screening and entered the study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population<br>(Selected Outputs) |
| All<br>Participants/Safet<br>y | <ul> <li>All participants who were randomized and received at least one dose of study medication.</li> <li>This population will be used for the study population and safety displays.</li> </ul> | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) | <ul> <li>Participants in the 'All Participants' population for whom a pharmacokinetic sample was obtained and had evaluable PK assay results.</li> <li>PK population will be the population for reporting of PK data.</li> </ul> | PK |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised in the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code Description | | Description | Order in TLF |
| Α | Prototype A | Prototype A | 1 |
| В | Prototype B | Prototype B | 2 |
| R | 2x5mg DTG Dispersible Tablets dispersed in water | DTG Ref | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Prototype A vs DTG Reference Treatment
- 2. Prototype B vs DTG Reference Treatment

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the last pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments Considered as Baseline | | | Baseline Used in |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Vital Signs | | Х | | Day -1 |
| Clinical Laboratory | | X | | Day -1 |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "All Participants" population, unless otherwise specified. Screen failures will be summarised or listed based on the "Screened" population.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

## 6.2. Details of Planned Study Population Summaries

### **Participant Disposition**

#### Participant Disposition for the Subject Conclusion Record

The number and percentage of participants who completed the study as well as participants who withdrew from the study will be summarized. Reason for withdrawal will also be summarized for participants who withdrew from the study. Only the total column will appear.

## Treatment Status and Reasons for Discontinuation of Study Treatment

A summary of the number and percentage of subjects who completed the study treatment as planned as well as subjects who stopped study treatment prematurely will be produced. Only the total column will appear.

#### Screening Status and Reasons for Screen Failure

This will be based on Screened population. The number and percentage of subjects who passed screening and who failed screening will be summarized along with the reasons for screen failure. Only the total column will appear.

#### Number of Subjects Enrolled by Country and Site ID

This will be based on Enrolled population. The number of subjects summarized by Country, Site ID and Investigator name will be presented. Only the total column will appear.

#### **Protocol Deviations**

#### Important Protocol Deviations

The number and percentage of subjects who had important protocol deviations defined as part of the protocol deviation management plan for the study, will be summarized. Only the total column will appear.

## **Demographic and Baseline Characteristics**

#### Demographic Characteristics

The number and percentage of subjects or summary statistics will be provided for each demographic characteristic and only the total column will appear: Sex, Age (years), Age Group (years), Ethnicity, Race detail, Height, Weight, and Body Mass Index. Age Group (years) will be categorized into three ('≤18', '19-55', '≥56'). Each demographic characteristic will be summarized using the minimum set of summary statistics.

#### Age Ranges

This will be based on Enrolled population. The number and percentage of subjects within each age range category will be provided. Only the total column will appear. Only age ranges that are applicable to the study will be included (i.e., only '18-55 years'). This is based on the standard of EMA clinical trial results disclosure requirements.

#### Race and Racial Combinations

The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. Only the total column will appear.

#### **Prior and Concomitant Medications**

All prior and concomitant medications will be summarized based on the definition specified in Appendix 3 later in the document.

## 7. SAFETY ANALYSES

The safety analyses will be based on the "All Participants" population, unless otherwise specified. No formal statistical analysis of the safety data will be conducted.

Unless stated otherwise, descriptive summaries for continuous variables will include n, mean, standard deviation (SD), median, minimum, maximum; whereas, n and percent will be used as summary statistics for categorical variable.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. Tables will present AEs in the treatment phase. Listings will present all AEs. The details of the planned displays are provided in Appendix 9: List of Data Displays.

#### 7.1.1. Details of Planned Adverse Event Summaries

Summaries will be provided by Period (Prototype A, Prototype B, DTG Reference Treatment) unless otherwise specified.

#### **Adverse Events (AEs)**

#### All AEs by SOC and PT

The number and percentage of subjects with all relevant adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### All AEs by Maximum Grade by SOC and PT

The number and percentage of subjects with adverse events by grade will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Drug-related AEs by SOC and PT

The number and percentage of subjects with all drug-related adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Drug-related AEs by Maximum Grade by SOC and PT

The number and percentage of subjects with drug-related adverse events by grade will be summarized by MedDRA System Organ Class and Preferred Term by treatment group

and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Common AEs

Summaries of the number and percentage of subjects with common (incidence greater than five percent) adverse events by overall frequency will be displayed for grade 2-4 events, non-serious events by SOC and PT, and drug related grade 2-4 events. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### **Serious Adverse Events**

#### Serious AEs by SOC and PT

The number and percentage of subjects with serious adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. All laboratory data will be summarized and listed. The details of the planned displays are in Appendix 9: List of Data Displays.

## 7.2.1. Details of Planned Laboratory Summaries

### Changes from Baseline

Changes in value from baseline for each quantitative laboratory test will be summarised at every assessed time point using descriptive statistics defined above.

#### Worst Case Laboratory Results by PCI Criteria Post-Baseline Relative to Baseline

The number of subjects with worst case laboratory results relative potential clinical importance (PCI) criteria which are post-baseline relative to baseline will be summarized by laboratory test and category.

#### Laboratory Results by Maximum Grade Increases Post-Baseline Relative to Baseline

The number of subjects with laboratory results will be summarized by laboratory test, term (e.g. CTCAE term), maximum grade increase (e.g., Increase to Grade 1, Increase to Grade 2, Increase to Grade 3, Increase to Grade 4) and maximum grade increase subtotals (e.g., Increase to Grades 1 to 4, Increase to Grades 2 to 4, Increase to Grades 3 to 4). Hepatobiliary results will also be summarized.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. Change from baseline in vital signs will be summarized descriptively. All ECG and vital signs data will be listed. The details of the planned displays are presented in Appendix 9: List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES

## 8.1. Primary Pharmacokinetic Analyses

## 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters of DTG will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC <sub>(0-t)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| AUC <sub>(0-inf)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC <sub>(0-inf)</sub> ) will be calculated as follows: $AUC_{(0-inf)} = AUC_{(0-inf)} + C_t / \lambda_z$ |
| C <sub>max</sub> (ng/mL) | Maximum observed plasma concentration following each dose will be obtained directly from the concentration-time data. |

#### NOTES:

- Additional parameters may be included as required.
- C<sub>t</sub> is the last observed quantifiable concentration.
- $\lambda_z$  is the first order rate constant associated with the terminal (log-linear) portion of the curve.

## 8.1.2. Summary Measure

The ratio of geometric means for  $AUC_{(0-t)}$ ,  $AUC_{(0-inf)}$  and  $C_{max}$  of DTG between each of the prototypes and DTG reference treatment will be used for the comparison between Prototype A vs. DTG Reference Treatment, and Prototype B vs. DTG Reference Treatment.

#### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events which may affect the evaluation of bioequivalence and food effect are not anticipated.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

#### 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

Derived PK parameters of DTG:

- AUC<sub>(0-t)</sub>
- AUC<sub>(0-inf)</sub>
- C<sub>max</sub>

#### **Model Specification**

 To evaluate the relative bioavailability of equivalent doses of single dose prototype liquid formulations containing 10mg equivalent DTG (Prototypes A and B) compared to a single dose of 2 x 5mg dispersible DTG tablet dispersed in water (DTG Reference Treatment), the PK parameters will be analysed using a mixed effect model as described below:

$$log_e$$
 (PK parameter) =  $\beta_0 + \gamma_i + \tau_j + \epsilon_{ij}$ 

where,

Bo: intercept

 $\gamma_i$ : random effect for ith participant, following N(0,  $\sigma_b^2$ )

τ<sub>i</sub>: treatment effect (j = Prototype A or Prototype B or DTG Reference Treatment)

 $\epsilon_{ij}$ : random error for participant i, treatment effect j, following N(0,  $\sigma_w^2$ ).

- The model parameters will be estimated using Restricted Maximum Likelihood with the Newton-Raphson algorithm.
- The Kenward-Roger degree of freedom approach will be used.
- Given the random effect for subject "i", the random error is assumed to be independently distributed within the subject.
- The least square means for each treatment formulation (Prototype A, Prototype B and DTG Reference Treatment) will be estimated based on the fitted model. The mean difference between the treatment formulations (Prototype A vs. DTG Reference Treatment, and Prototype B vs. DTG Reference Treatment) and its 90% CIs will be also estimated using the withinsubject variance.
- The estimates of least square means for each treatment formulation, the treatment difference between treatment formulations and the 90% CIs will be exponentially back-transformed to obtain the estimates of geometric means of AUC<sub>(0-t)</sub>, AUC<sub>(0-t)</sub>, and C<sub>max</sub> for each treatment

formulation, the ratio of geometric means (Prototype A/DTG Reference, Prototype B/DTG Reference) and its 90% CIs, respectively.

 Within-subject variability (%CVw) for the PK parameters will be estimated using within-subject variance from the analysis model as follows:

%CVw (%) = 
$$[\exp(\sigma_w^2) - 1]^{1/2}$$
 x 100

#### **Model Checking & Diagnostics**

In case there is a problem with model convergence, the arithmetic means for loge-transformed AUC<sub>(0-t)</sub> and C<sub>max</sub> and the treatment differences (Prototype A vs. DTG Reference, Prototype B vs. DTG Reference) within each participant will be calculated using only data from the participants who have completed both the periods for Prototype A and DTG Reference (and Prototype B and DTG Reference, for the second comparison). The mean treatment difference and paired-t test based 90% CIs for treatment difference in loge scale will be estimated. The results will be provided in an exponentially back-transformed scale.

#### **Model Results Presentation**

Based on the relative bioavailability, the bioequivalence between Prototypes A, B and DTG Reference Treatment will be evaluated as follows:

- The bioequivalence is established when the 90% CI of the ratio for AUC<sub>(0-t)</sub>, AUC<sub>(0-inf)</sub> and C<sub>max</sub> between treatment formulations (Prototype A vs. DTG Reference Treatment, and Prototype B vs. DTG Reference Treatment) are within the range of 0.80 to 1.25.
- Even if the 90% CI doesn't meet the above criteria, the bioequivalence is established when the point estimate of the ratio for AUC<sub>(0-t)</sub>, AUC<sub>(0-inf)</sub> and C<sub>max</sub> between treatment formulations are within the range of 0.90 to 1.11.

#### 8.1.6. Details of Planned Pharmacokinetic Displays

Analysis of relative bioavailability of Prototypes A and B vs. DTG Reference Treatment for  $\underline{AUC}_{(0-i)}$ ,  $\underline{AUC}_{(0-inf)}$  and  $\underline{C}_{max}$ 

The analysis results will be presented as described in Section 8.1.5.1 - Model Results Presentation.

# 8.2. Secondary Pharmacokinetic Analyses

#### 8.2.1. Endpoint / Variables

#### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Standards for Pharmacokinetic)

#### 8.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters of DTG will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher. All calculations of non-compartmental parameters will be

based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC <sub>(0-t)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| AUC <sub>(0-inf)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC <sub>(0-inf)</sub> ) will be calculated as follows: $AUC_{(0-inf)} = AUC_{(0-t)} + C_t / \lambda_z$ |
| AUC <sub>(0-24)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) to 24 hours post-dose. |
| AUC <sub>(0-72)</sub><br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) to 72 hours post-dose. |
| C <sub>max</sub> (ng/mL) | Maximum observed plasma concentration following each dose will be obtained directly from the concentration-time data. |
| C <sub>24</sub> (ng/mL) | The observed concentration at 24h post-dose. |
| C <sub>t</sub> (ng/mL) | The last observed quantifiable concentration. |
| t <sub>max</sub> (h) | The time to maximum observed plasma drug concentration following each dose will be obtained directly from the concentration-time data. |
| t <sub>1/2</sub> (h) | Terminal half-life will be calculated as follows: $t_{1/2} = ln2 \ / \ \lambda_z$ |
| t <sub>lag</sub> (h) | Absorption lag time. |
| t (h) | The time of last quantifiable concentration. |
| %AUCex (%) | The percentage of AUC <sub>(0-inf)</sub> obtained by extrapolation (%AUCex) will be calculated as follows: %AUCex = (AUC <sub>(0-inf)</sub> – AUC <sub>(0-inf)</sub> / AUC <sub>(0-inf)</sub> x 100 |
| CL/F<br>(mL/h) | Apparent clearance following oral dosing will be calculated as follows: CL/F = Dose / AUC <sub>(0-inf)</sub> |
| Vz/F<br>(mL) | Apparent volume of distribution after oral administration will be calculated as follows: $Vz/F = Dose / (\lambda_z \times AUC_{(0-inf)})$ |
| λ <sub>z</sub> (/h) | The first order rate constant associated with the terminal (log-linear) portion of the curve. |

#### NOTES:

Additional parameters may be included as required.

## 8.2.2. Summary Measure

Descriptive summaries of the above defined parameters except  $t_{max}$  will be presented. Unless stated otherwise, descriptive summaries for continuous variables will include n, mean, standard deviation (SD), median, minimum, maximum; whereas, n and percent will be used as summary statistics for categorical variable. Geometric mean with

associated 95% CI, and the between-subject coefficient of variance (CV) (%CVb) for the geometric mean will be included for PK variables, where applicable.

For the t<sub>max</sub>, point estimates and associated 90% confidence intervals for the median differences between treatment formulations (Prototype A, Prototype B) and DTG Reference Treatment will be presented.

#### 8.2.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events which may affect the evaluation of bioequivalence and food effect are not anticipated.

## 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.2.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

t<sub>max</sub>

#### **Model Specification**

 A non-parametric analysis of this endpoint will be performed by using Wilcoxon matched pair test.

#### **Model Results Presentation**

 Point estimates and associated 90% confidence intervals for the median differences between treatment formulations (Prototypes A and B) and DTG Reference Treatment will be presented.

#### 8.2.6. Details of Planned Pharmacokinetic Displays

Summaries will be provided by treatment formulations (Prototype A, Prototype B and DTG Reference Treatment), unless otherwise specified.

#### DTG Plasma Concentration-Time Data

DTG plasma concentrations at every scheduled time point will be summarized using n, mean, standard deviation, median, minimum, and maximum.

#### Derived DTG Plasma Pharmacokinetic Parameters (non-transformed)

DTG plasma pharmacokinetic parameters defined in Section 8.2.1 will be summarized using n, mean, 95% CI, standard deviation, median, minimum, and maximum.

### Derived DTG Plasma Pharmacokinetic Parameters (log-transformed)

For each pharmacokinetic parameter with a log-normal distribution (AUC<sub>(0-t)</sub>, AUC<sub>(0-inf)</sub>,  $C_{max}$ ,  $t_{1/2}$ , %AUCex, CL/F, Vz/F,  $\lambda_z$ ), the log-transformed parameters will be summarized using n, geometric mean, 95% CI of geometric mean, standard deviation of log-transformed data and between subject coefficient of variation (%CVb).

#### Non-Parametric Analysis of the Pharmacokinetic Parameter $t_{max}$

For  $t_{max}$ , point estimates of the treatment differences in median along with its 90% CI will be presented. Also, the individual estimates of median of each treatment formulations (Prototypes A and B) and DTG Reference Treatment will be presented along with the n of each group.

# 9. REFERENCES

GlaxoSmithKline Document Number 2018N379348\_01 Study ID 209354. A non-randomized, sequential, fixed-sequence evaluation of prototype dolutegravir liquid formulations versus 5mg dolutegravir dispersible tablets following single-dose fasted-state administrations to normal healthy adult participants. 2019.

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Not applicable, as there is no Per Protocol Population defined for this study.

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

## 10.2.1.1. Screening Assessments

| Visit Window (relative to Day 1) | Day -30<br>to -2 | Notes |
|---|---|---|
| Informed Consent | Χ | |
| Demographics | Χ | |
| Physical examination height, weight and BMI | Χ | |
| Medical/medication/ history | Х | Medical/medication/drug and alcohol history will be recorded at screening and updated at admission. |
| Urine drug / Cotinine and Breathalyzer screening | Х | |
| 12-lead ECG and Vital Signs | Х | |
| Serum or urine hCG test (female participants only) | Х | <ul> <li>See inclusion criterion for female participants.</li> <li>Performed at site standard procedure.</li> </ul> |
| FSH and estradiol (women) | Χ | |
| HIV, Hep B and Hep C Screen | Х | |
| Hematology/Chemistry/Urinalysis tests | Х | |

BMI: Body mass index, ECG: Electrocardiogram, hCG: Human chorionic gonadotropin, FSH: Follicle stimulating hormone; HIV: Human immunodeficiency virus, Hep B: Hepatitis B; Hep C: Hepatitis C

#### 10.2.1.2. Treatment Period Assessments

| | All Dosing Periods | | | | | | | | Notes • Day -1 of Periods 2 and 3 may be the same day as Day 6 |
|---|---|---|---|---|---|---|---|---|---|
| | | Day 1 | | | Day 2 | Day 3 | Day 4 | Day 4 💂 | of prior periods |
| Assessments | Day -<br>1 | Pre-<br>dose | 0<br>hr | Post Dose | - | 48 hr | 72 hr | Follow-up | <ul> <li>At Follow-up – Participants with no ongoing AEs or Vital Sign/Laboratory measures of clinical concern may be followed virtually by the site via telephone contact.</li> <li>Follow-up assessments should be completed in the event of an early participant termination.</li> </ul> |
| Admission to Unit | Χ | | | | | | | | |
| Discharge | | | | | | Χ | | | |
| Outpatient Visit | | | | | | | Х | Х | Follow-up visit will occur 7 to 14days post last dose. |
| 12-lead ECG | Х | | | | | | | | Single ECGs will be collected at Screening and on Day-1 of Period 1 only. Additional ECGs may be performed at the discretion of the investigator. |
| Vital signs | Χ | | | | | | Χ | Χ | Single measurements performed at all time points. |
| Brief Physical Exam | X | | | | | | | | Brief examinations may be made full examinations and |
| Urine Drug / Cotinine and Breathalyzer | Х | | | | | | | | laboratory procedures may be repeated, if needed, at the discretion of the Investigator. |
| Clinical laboratory tests | Х | | | | | | | X* | <ul> <li>Illicit Drug/Alcohol/Cotinine screening will be performed in accordance with the sites' standard practice.</li> <li>Clinical laboratory tests – see Table 6 of Study Protocol.</li> <li>*Clinical laboratory tests at follow-up are only necessary if participant had a previous abnormal lab value</li> </ul> |
| Dosing | | | Х | | | | | | Participant will be dosed while in the seated position. |
| Meals | Χ | | | Post 4-hour PK sample | Pe | r standar | at the cli | nic | Participants will fast from 10hrs pre-dose to 4-hours post-dose. |
| Pharmacokinetic Sampling | | Х | | Collect at 0.25, 0.5, 0.75<br>3.5, 4, 5, 6, 8, 12, 16, 2<br>post-dos | 24, and 48-hours X | | Х | | <ul> <li>Pre-dose (within 15 minutes prior to dosing).</li> <li>4-hour post dose sample must be taken <u>prior to</u> provision of food.</li> <li>Permitted window for the collection of PK sample at each time point is specified in Section 8.5.1. of Study Protocol.</li> </ul> |
| Adverse Events/SAEs | Х | <b>←===</b> | <b>←</b> ======X======X======================= | | | ====→ | Х | | |
| Concomitant medications | Х | <b>←===</b> : | X | | | <b>&gt;</b> | Х | | |

# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 10.3.1. Study Phases

Assessments and events (e.g., study withdrawal) will be classified according to the time of occurrence relative to dosing start Date and Time by Period.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Reference Day ≤ Previous Day of Dosing Start Date in Period 1 |
| Period 1 | Previous Day of Dosing Start Date in Period 1 < Reference Day ≤ Previous Day of Dosing Start Date in Period 2 |
| Period 2 | Previous Day of Dosing Start Date in Period 2 < Reference Day $\leq$ Previous Day of Dosing Start Date in Period 3 |
| Period 3 | Previous Day of Dosing Start Date in Period 3 < Reference Day ≤ Dosing Start Date in Period 3 + 4 Days |
| Post-Treatment | Reference Day > Dosing Start Date in Period 3 + 4 Days |

# 10.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 7 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.3.2. Treatment Emergent Flag for Adverse Events

| Study Phase | Definition |
|---|---|
| Pre-Treatment | AE Onset Date and Time < Study First Dosing Start Date and Time |
| Period 1 | Study First Dosing Start Date and Time $\leq$ AE Onset Date and Time $<$ Dosing Start Date and Time in Period 2 |
| Period 2 | Dosing Start Date and Time in Period 2 $\leq$ AE Onset Date and Time $<$ Dosing Start Date and Time in Period 3 |
| Period 3 | Dosing Start Date and Time in Period $3 \le$ AE Onset Date and Time $\le$ Dosing Start Date and Time in Period $3 + 4$ Days |
| Post-Treatment | AE Onset Date and Time > Dosing Start Date in Period 3 + 4 Days |
| Time since Study | If study phase of the event is pre-treatment, |
| First Dose (min) | AE Onset Date and Time - Study First Dosing Start Date and Time |
| | otherwise |
| | AE Onset Date and Time – Study First Dosing Start Date and Time + 1 min |
| Time since Period | If study phase of the AE is Pre-Treatment, set to missing |
| First Dose (min) | If study phase of the AE is Period 1, |
| | AE Onset Date and Time – Dosing Start Date and Time in Period 1 + 1 min |
| | If study phase of the AE is Period 2, |
| | AE Onset Date and Time – Dosing Start Date and Time in Period 2 + 1 min |
| | If study phase of the AE is Period 3, |
| | AE Onset Date and Time – Dosing Start Date and Time in Period 3 + 1 min |
| | If study phase of the AE is Post-Treatment, |
| | AE Onset Date and Time – (Dosing Start Date in Period 3 + 4 Days) + 1 min |
| Duration (min) | AE Resolution Date and Time – AE Onset Date and Time + 1 min |
| Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be treatment emergent.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

## 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software 9.4 will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound | : \ARPROD\GSK1349572\MID209354\ |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1].</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated. | |

# 10.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | | |
|---|---|---|
| | Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |

| Categorical Data | N, n, frequency, % |
|---|---|
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487 Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | Pharmacokinetic Parameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | No PK parameters derived by programmer are planned |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters in GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards: Standards for the Transfer and Reporting of PK Data using HARP |

## 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### **Period Day**

- Calculated as the number of days from Dosing Date in Period 1 or Period 2 or Period 3.
  - If Study Phase of Ref Assessment or Event = Pre-Treatment or Missing
    - → Period Day = Missing
  - If Study Phase of Ref Assessment or Event = Period 1
    - → If Ref Date is on or after Dosing Date in Period 1, Period Day = Ref Date Dosing Date in Period 1 + 1 day
  - If Study Phase of Ref Assessment or Event = Period 2
    - → If Ref Date is on or after Dosing Date in Period 2, Period Day = Ref Date Dosing Date in Period 2 + 1 day
  - If Study Phase of Ref Assessment or Event = Period 3
    - → If Ref Date is on or after Dosing Date in Period 3, Period Day = Ref Date Dosing Date in Period 2 + 1 day
  - If Study Phase of Ref Assessment or Event = Post-Treatment
    - $\rightarrow$  If Ref Date is after Dosing Date in Period 3 + 4 Days, Period Day = Ref Date (Dosing Date in Period 3 + 4 Days) + 1 day

## 10.5.2. Study Population

#### **Extent of Exposure**

- Number of days of exposure to study drug for each period will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were enrolled but did not report a treatment start date will be categorised as having zero days of exposure.

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - A date and month will be imputed as '30th June' as it will not be captured.
- Date of Informed Consent will be used as reference date of calculation.

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study including the follow up visit.</li> <li>Withdrawn participants may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF does not allow for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month will not be missing.</li> <li>The eCRF allows for the possibility of missing times to be recorded for AE start and end</li> </ul> |
| | dates. Missing times will be imputed using the following convention: |
| | o If the missing time is a start time, a '00:00' will be used for the time. |
| | o If the missing time is a stop time, a '23:59' will be used for the time. |
| | The recorded missing time will be displayed in listings without imputed values. |
| Concomitant<br>Medications/<br>Medical | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be</li> </ul> |
| History | used for the month |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent<br/>on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | <ul> <li>The eCRF allows for the possibility of missing times to be recorded for concomitant<br/>medications start and end dates. Missing times will be imputed using the following<br/>convention:</li> </ul> |
| | <ul> <li>If the missing time is a start time, a '00:00' will be used for the time.</li> </ul> |
| | <ul> <li>If the missing time is a stop time, a '23:59' will be used for the time.</li> </ul> |
| | The recorded partial date and missing time will be displayed in listings without imputed values. |

# 10.7. Appendix 7: Values of Potential Clinical Importance

Any DAIDS Grade 2 or above event will be treated as an event of potential clinical importance.

Please refer to the link below for more details:

https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf

# 10.8. Appendix 8: Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | |
| CDISC | Analysis and Reporting |
| CI | Clinical Data Interchange Standards Consortium Confidence Interval |
| CPMS | |
| | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTC | Common Terminology Criteria for Adverse Events |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| 1 1/ 11/11/00 | Kandomization & Medication Ordering System |

| Abbreviation | Description |
|--------------|---------------------------------|
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TMF | Trial Master File |

# 10.8.2. Trademarks

| Trademarks of the ViiV Healthcare Group of Companies |
|------------------------------------------------------|
| None |

| Trademarks not owned by the ViiV<br>Healthcare Group of Companies |
|-------------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.9. Appendix 9: List of Data Displays

# 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|----------------|
| Study Population | 1.1 to 1.12 | Not Applicable |
| Safety | 3.1 to 3.21 | Not Applicable |
| Pharmacokinetic | 4.1 to 4.5 | 4.1 to 4.5 |
| Section | List | ings |
| ICH Listings | 1 to | 33 |

# 10.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------|--------|-------|----------------|
| Pharmacokinetic | PK_Fn | PK_Tn | Not Applicable |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |
# 10.9.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | All<br>Participants | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | Only "Total" column will appear Please refer to mock shell DM1 in Appendix 10 for an idea of how a typical study population display would look like. | SAC |
| 1.2. | All<br>Participants | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | Only "Total" column will appear | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Only "Total" column will appear | SAC |
| 1.4. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | Only "Total" column will appear | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | All<br>Participants | DV1 | Summary of Important Protocol Deviations | Only "Total" column will appear | SAC |
| Popula | tion Analysed | | | | |
| 1.6. | Enrolled | SP1 | Summary of Study Populations | | SAC |
| Demog | raphic and Bas | seline Characteris | tics | 1 | 1 |
| 1.7. | All<br>Participants | DM3 | Summary of Demographic Characteristics | Only "Total" column will appear | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Enrolled | DM11 | Summary of Age Ranges | Only "Total" column will appear | SAC |
| 1.9. | All<br>Participants | DM5 | Summary of Race and Racial Combinations | Only "Total" column will appear | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 1.10. | All<br>Participants | MH1 | Summary of Past Medical Conditions | Only "Total" column will appear | SAC |
| 1.11. | All<br>Participants | MH1 | Summary of Current Medical Conditions | Only "Total" column will appear | SAC |
| 1.12. | All<br>Participants | CM1 | Summary of Concomitant Medications | Only "Total" column will appear | SAC |

# 10.9.5. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | All<br>Participants | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | Include "Total" column Please refer to mock shell AE1CP in Appendix 10 for an idea of how a typical safety display would look like. | SAC |
| 3.2. | All<br>Participants | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term | Include "Total" column | SAC |
| 3.3. | All<br>Participants | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | Include "Total" column | SAC |
| 3.4. | All<br>Participants | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | Include "Total" column | SAC |
| 3.5. | All<br>Participants | AE1CP | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | Include "Total" column | SAC |
| 3.6. | All<br>Participants | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade | Include "Total" column | SAC |
| 3.7. | All<br>Participants | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | Include "Total" column | SAC |
| 3.8. | All<br>Participants | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency | Include "Total" column | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 3.9. | All<br>Participants | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | Include "Total" column | SAC |
| Labora | tory: Chemistry | / | | | |
| 3.10. | All<br>Participants | LB1 | Summary of Chemistry Changes from Baseline | Include "Total" column | SAC |
| 3.11. | All<br>Participants | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | Include "Total" column | SAC |
| 3.12. | All<br>Participants | LB16 | Summary of Worst Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | Include "Total" column | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.13. | All<br>Participants | LB1 | Summary of Hematology Changes from Baseline | Include "Total" column | SAC |
| 3.14. | All<br>Participants | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | Include "Total" column | SAC |
| 3.15. | All<br>Participants | LB16 | Summary of Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | Include "Total" column | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | |
| 3.16. | All<br>Participants | LB1 | Summary of Urine Concentration Changes from Baseline | Include "Total" column | SAC |
| 3.17. | All<br>Participants | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | Include "Total" column | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborat | tory: Hepatobil | iary (Liver) | | | |
| 3.18. | All<br>Participants | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | Include "Total" column | SAC |
| 3.19. | All<br>Participants | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | Include "Total" column | SAC |
| Vital Sig | gns | | | | |
| 3.20. | All<br>Participants | VS1 | Summary of Change from Baseline in Vital Signs | Only "Total" column will appear | SAC |
| 3.21. | All<br>Participants | VS3 | Summary of Worst Case Vital Signs Results by Maximum Grade Increase Post-Baseline Relative to Baseline | Only "Total" column will appear | SAC |

#### 10.9.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1. | PK | PK01 | Summary of DTG Plasma Concentration-Time Data | | SAC |
| 4.2. | PK | PK03 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (non-transformed) | | SAC |
| 4.3. | PK | PK05 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (log-transformed) | | SAC |
| 4.4. | PK | PK_T1 | Non-parametric Analysis of tmax | Refer to example shell | SAC |
| 4.5. | PK | PK_T2 | Analysis of Relative Bioavailability of Prototype Formulations vs. DTG Reference Treatment for Cmax, AUC(0-t), and AUC(0-inf) | Refer to example shell | SAC |

# 10.9.7. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1. | PK | PK16b | Individual DTG Plasma Concentration-Time Plots by Participant | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 4.2. | PK | PK16b | Individual DTG Plasma Concentration-Time Plots by Treatment | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 4.3. | PK | PK17 | Mean (+SD) DTG Plasma Concentration-Time Plots | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 4.4. | PK | PK18 | Median DTG Plasma Concentration-Time Plots | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 4.5. | PK | PK_F1 | Plot of Individual DTG Plasma Cmax, AUC(0-t), and AUC(0-inf) by Treatment | Refer to example shell | SAC |

# 10.9.8. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | · |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All<br>Participants | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | All<br>Participants | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | All<br>Participants | TA2 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 5. | All<br>Participants | DV2A | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 6. | All<br>Participants | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | • |
| 7. | All<br>Participants | SP3a | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | · | |
| 8. | All<br>Participants | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 9. | All<br>Participants | DM10 | Listing of Race | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 10. | All<br>Participants | CM5 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 11. | All<br>Participants | EX4 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | - | |
| 12. | All<br>Participants | AE9CP | Listing of All Adverse Events | ICH E3 | SAC |
| 13. | All<br>Participants | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 14. | All<br>Participants | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 15. | All<br>Participants | AE9CPa | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 16. | All<br>Participants | AE9CPa | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 17. | All<br>Participants | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 18. | All<br>Participants | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| 19. | All<br>Participants | AE8 / AECP8 /<br>AE9 / AE9CP | Listing of Other Significant Adverse Events | ICH E3 | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hepato | biliary (Liver) | | | | |
| 20. | All<br>Participants | MH3 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 21. | All<br>Participants | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |
| All Lab | oratory | | | | |
| 22. | All<br>Participants | LB6 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 23. | All<br>Participants | LB6 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 24. | All<br>Participants | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 25. | All<br>Participants | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 26. | All<br>Participants | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 27. | All<br>Participants | EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 28. | All<br>Participants | EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| 29. | All<br>Participants | EG6 | Listing of Abnormal ECG Findings | IDSL | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | gns | | | | |
| 30. | All<br>Participants | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 31. | All<br>Participants | VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |
| PK | | | | | |
| 32. | All<br>Participants | PK08 | Listing of DTG Plasma Pharmacokinetic Concentration-Time Data | IDSL | SAC |
| 33. | All<br>Participants | PK14 | Listing of Derived DTG Plasma Pharmacokinetic Parameters | IDSL | SAC |

#### 10.10. Appendix 10: Example Mock Shells for Data Displays

Example DM1

Protocol: 209354 Page 1 of 3

Population: All Patients

Table X Summary of Demographic Characteristics

| | Total |
|---------------------|-----------|
| | (N=200) |
| Sex | |
| n | 200 |
| F | 100 (50%) |
| M | 100 (50%) |
| Age (YEARS)[1] | |
| n | 200 |
| Mean | 50.0 |
| SD | 10.00 |
| Median | 50.0 |
| Min. | 18 |
| Max. | 65 |
| Age Group(YEARS)[1] | |
| <=18 | 5 (3%) |
| 19-64 | 100 (50%) |
| >=65 | 95 (48%) |

<sup>[1]</sup> Age is imputed when full date of birth is not provided.

### Example AE1CP

Protocol: 209354 Page 1 of n

Population: All Patients

| System Organ Class<br>Preferred Term | Prototype A | Prototype B (N=78) | DTG Reference T | Total<br>N=78) |
|---|---|---|---|---|
| ANY EVENT | 58 (74%) | 64 (82%) | 64 (85%) 65 | (83%) |
| Gastrointestinal disorders Any event Dyspepsia Nausea Vomiting Nos Constipation Diarrhoea Nos Toothache Abdominal Pain Upper Dry Mouth Flatulence Gastrointestinal Upset Haemorrhoids Salivary Hypersecretion Abdominal Tenderness Hyperacidity Loose Stools Abdominal Pain Nos Faecal Incontinence Gastritis Nos Lip Disorder Nos Lip Dry Stomach Discomfort | 28 (36%<br>9 (12%<br>6 (8%<br>3 (4%)<br>6 (8%)<br>2 (3%)<br>3 (4%)<br>1 (1%)<br>0<br>1 (1%)<br>0<br>0<br>0<br>0<br>1 (1%)<br>0<br>0<br>0<br>0<br>0<br>0<br>0 | 11 (14%) 8 (10%) 10 (13%) 6 (8%) 4 (5%) 1 (1%) 2 (3%) 1 (1%) 3 (4%) 1 (1%) 0 2 (3%) 2 (3%) 1 (1%) 2 (3%) | 5 (7%) 15<br>4 (5%) 11<br>3 (4%) 7<br>2 (3%) 6<br>3 (4%) 5<br>2 (3%) 5<br>4 (5%) 5<br>1 (1%) 4<br>3 (4%) 3<br>0 3<br>1 (1%) 2<br>0 2<br>1 (1%) 2<br>0 2<br>1 (1%) 2<br>1 (1%) 2<br>1 (1%) 1 | (8%)<br>(6%)<br>(6%)<br>(5%)<br>(4%)<br>(3%)<br>(3%)<br>(3%)<br>(1%)<br>(1%)<br>(1%)<br>(1%) |
| Nervous system disorders<br>Any event<br>Headache<br>Dizziness<br>Extrapyramidal Disorder | 28 (36%,<br>15 (19%,<br>3 (4%,<br>4 (5%, | 11 (14%)<br>8 (10%) | 14 (19%) 27 3 (4%) 11 | , , |

Example: PK T1 Page 1 of n

Protocol: 209354 Population: PK

Table X

Analysis of Relative Bioavailability of Prototype Formulations vs. DTG Reference Treatment fo

Analysis of Relative Bioavailability of Prototype Formulations vs. DTG Reference Treatment for Cmax, AUC(0-t), and AUC(0-inf)

| Parameter | Treatment<br>Comparison | | Adjusted | Geom | Mean | Ratio<br>(trt2/trt1) | 90% CI | %CVw[1] |
|---|---|---|---|---|---|---|---|---|
| rarameter | Comparison | n | Test | n | Ref | _ (6162/6161) | 300 01 | 00 V W [1] |
| Cmax (unit) | trt1 vs<br>ref | XX | xx.xxx | XX | xx.xx | x.xxx | (x.xxx, x.xxx) | x.xxx |
| ( ) | trt2 vs<br>ref | XX | XX.XXX | XX | XX.XXX | x.xxx | (x.xxx, x.xxx) | x.xxx |
| AUC(0-t)(unit) | trt1 vs<br>ref | XX | xx.xxx | XX | xx.xxx | x.xxx | (x.xxx, x.xxx) | x.xxx |
| | trt2 vs<br>ref | XX | xx.xxx | XX | xx.xxx | x.xxx | (x.xxx, x.xxx) | x.xxx |
| AUC(0-inf) (unit) | trt1 vs<br>ref | XX | XX.XXX | XX | xx.xxx | x.xxx | (x.xxx, x.xxx) | x.xxx |
| | trt2 vs<br>ref | XX | xx.xxx | XX | xx.xxx | x.xxx | (x.xxx, x.xxx) | x.xxx |

[1] Within-subject variability of each PK parameter

trt1 = "Prototype A", trt2 = "Prototype B" trt3 = "DTG Reference"

#### CONFIDENTIAL

209354

Example: PK\_F1 Page 1 of n

Protocol: 209354
Population: PK



Note: Geometric mean and 95% CI

#### Programming notes:

Add three treatments - trt1 = "Prototype A", trt2 = "Prototype B" trt3 = "DTG Reference" Figures will be presented in left (Cmax), center (AUC(0-t), and right (AUC(0-inf).